CLINICAL TRIAL: NCT02000765
Title: An Open-Label, Non-Randomized, Two-Period, Cross-Over, Mass Balance Study to Investigate the Recovery, Excretion and Pharmacokinetics of 14C-GSK2140944 Administered as a Single Intravenous and Single Oral Dose to Healthy Adult Male Subjects (BTZ115774)
Brief Title: A Study to Investigate the Recovery, Excretion and Pharmacokinetics of [14C]-GSK2140944 Administered as a Single Intravenous and Single Oral Dose to Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115774
Record Dates: First submitted 2013-11-07; First posted 2013-12-04 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Infections, Respiratory Tract
Keywords: oral; ADME; IV; antibiotic; healthy volunteer; [14C]-GSK2140944; mass balance; radiolabel
MeSH Terms: conditions — Respiratory Tract Infections | interventions — gepotidacin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2140944 for Injection and Capsule (Experimental): Each subject will receive a single 1000 milligram (mg) IV dose of GSK2140944 containing [14C]-GSK2140944 of approximately 22.5 microcurie [μCi] (approximately 0.8 megabecquerel [MBq]) of radioactivity given as a 2 hour infusion on Day 1 of treatment period 1 and 2000 mg oral dose of GSK2140944 containing [14C]-GSK2140944 of approximately 45 μCi (approximately 1.7 MBq) of radioactivity on Day 1 of treatment period 2. Each treatment period will be followed with washout of atleast 8 Days.
  Interventions: Drug: GSK2140944 for Injection; Drug: GSK2140944 Capsule

INTERVENTIONS:
Drug: GSK2140944 for Injection — GSK2140944 (1 gram) for Injection will be supplied as powder for injection containing [14C] GSK2140944. Non sterile powder is to be dissolved aseptically in sterile water for injection to a concentration of 4 mg/mL free base equivalent. IV solution is prepared by sterile filtration. 250 mL of IV solution, equivalent to 1000 mg GSK2140944, is then administered intravenously.
Drug: GSK2140944 Capsule — GSK2140944 Capsule (2 gram) will be supplied as powder in capsule containing [14C] GSK2140944. Powder is to be filled in empty capsule to achieve 200-400 mg strength per capsules as free base equivalent. Sufficient capsules are administered to provide the required total dose of 2 gram as free base.

SUMMARY:
This is an open-label, non-randomized, two-period, cross-over, mass balance study that will evaluate the recovery, excretion, and pharmacokinetics of a single intravenous (IV) dose of [14C]-GSK2140944 (Period 1) and a single oral dose of [14C]-GSK2140944 ( Period 2) in 6 healthy male subjects. The results from this study will aid in the design of future clinical pharmacology studies such as the thorough corrected QT interval study, special population studies (renal, hepatic, critically ill patients), potential drug interaction studies, and will help to establish safe and efficacious intravenous and oral dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Male aged between 30 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter outside the reference range for the population being studied may be included only if the Investigator feels and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram and Body Mass Index within the range 19- 31 kilogram per square meter (inclusive).
* Alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* A history of regular bowel movements (averaging one or more bowel movements per day).
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Protocol. This criterion must be followed from the time of the first dose of study medication until four months after the last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 ml) of beer, 1 glass (125 milliliter [mL]) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy must be excluded.
* History of sensitivity to quinolones including photosensitivity and tendon rupture.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening or positive test for Human Immunodeficiency Virus (HIV) antibody.
* A screening or Day -1 urinalysis positive for protein or glucose (greater than "1+" findings of protein or glucose).
* A serum creatinine value between screening and Day -1 visit that is increased by more than 0.2 milligrams per decilitre (or 15.25 micromole per liter) changes.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* Exclusion criteria for screening and baseline ECG (a single repeat is allowed for eligibility determination): Heart rate <40 and >100 beats per minute; PR Interval <120 and >220 milliseconds (msec); QRS duration <70 and >100 msec; QT duration corrected for heart rate by Bazett's formula (QTcB) or QT duration corrected for heart rate by Fridericia's formula (QTcF) interval >450 msec; Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization); Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block [second degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses> 3 seconds, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.
* Where participation in the study would result in donation of blood or blood products in excess of 500 millilitre (mL) within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Subjects who have received a total body radiation dose of greater than 5.0 millisievert (upper limit of World Health Organization category II) or exposure to significant radiation (e.g. serial x-ray or CT scans, barium meal etc) in the 12 months prior to this study.

* Any condition that could interfere with the accurate assessment and recovery of radioactivity [14C].
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months.
* Unwillingness to commit to avoid excessive exposure to sunlight (or exposure whilst on a tanning bed) which would cause a sunburn reaction from first dose up to and including discharge.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
GSK2140944 PK parameters following single IV or oral doses of [14C]-GSK2140944 | Pre-dose and post dose(0 minute [min], 15 min, 30 min, 60 min, 120 min, 2.5 hour[hr], 3 hr, 4 hr, 6 hr, 6.5 hr, 8 hr, 12 hr, 16 hr, 24 hr, 48 hr, 72hr, 96 hr, 120hr, 144 hr, 168 hr, 48 hr, 72 hr, 96 hr, 120 hr, 144 hr and 168 hr) of each treatment period
  From the plasma concentration-time and blood/plasma radioactivity concentration-time data, the following pharmacokinetic parameters will be determined, as data permit: maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve [AUC(0-t) and AUC(0-∞)], and apparent terminal phase half-life (t1/2). Systemic clearance (CL) and volume of distribution (Vdss) of GSK2140944 may be calculated for IV regimen only.
Total recovery of radioactivity in urine and feces following separate single IV and oral doses of [14C]-GSK2140944 | Pre-dose and post dose(0-6 hr, 6 12 hr, 12 24 hr, 48 hr, 72 hr, 96 hr, 120 hr, 144 hr, 168 hr, 48 hr, 72 hr, 96 hr, 120 hr, 144 hr and 168 hr) of each treatment period
  Total recovery of radioactivity in urine and feces is defined as a percentage of total radioactive dose in each interval and cumulatively.

SECONDARY OUTCOMES:
Number of subjects with adverse events (AE) | Up to 7 weeks
Safety and tolerability of GSK2140944 after single IV and oral doses as assessed by concomitant medications review | Up to 7 weeks
Safety and tolerability of GSK2140944 after single IV and oral doses as assessed by clinical laboratory tests | Day 1 and Day 8 of each treatment period
  clinical laboratory tests includes hematology, clinical chemistry, urinalysis
Safety and tolerability of GSK2140944 after single IV and oral doses as assessed by electrocardiogram (ECG) | Day 1 (Pre dose and 1 hr, 2 hr, 4 hr and 8 hr post dose)and Day 8 of each treatment period
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT interval (QTc) intervals.
Safety and tolerability of GSK2140944 after single IV and oral doses as assessed by vital signs | Day 1 (Pre dose and 1 hr, 2 hr, 4 hr and 8 hr post dose)and Day 8 of each treatment period
  Vital sign measurements to be measurement include systolic and diastolic blood pressure, pulse rate and temperature.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115774 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115774?search=study&study_ids=115774#rs
- Available data/document: Annotated Case Report Form: 115774 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115774 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115774 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115774 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115774 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115774 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115774 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register